CLINICAL TRIAL: NCT05664971
Title: A Phase Ib/II Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Initial Efficacy of Recombinant Humanized Anti-BTLA Monoclonal Antibody (JS004) Injection Combined With Toripalimab and With Standard Chemotherapy in Patients With Advanced Lung Cancer
Brief Title: JS004 Combined With Toripalimab and With Standard Chemotherapy Treat Patients With Advanced Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS004-007-Ib/II-LC
Record Dates: First submitted 2022-11-28; First posted 2022-12-27 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Advanced Lung Cancer
MeSH Terms: interventions — Injections; toripalimab; Docetaxel; Pemetrexed; Cisplatin; Carboplatin; Paclitaxel; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): NSCLC-squamous carcinoma third line;JS004 200mg + JS001 240mg Q3w, maintained until disease progression
  Interventions: Biological: Recombinant humanized anti-BTLA monoclonal antibody (JS004) injection; Biological: Toripalimab
- Cohort 2 (Experimental): NSCLC-squamous carcinoma second line;JS004 200mg + JS001 240 mg + docetaxel Q3w, maintained until disease progression
  Interventions: Biological: Recombinant humanized anti-BTLA monoclonal antibody (JS004) injection; Biological: Toripalimab; Drug: Docetaxel
- Cohort 3 (Experimental): NSCLC-non-squamous carcinoma first line;JS004 200mg + JS001 240 mg + pemetrexed + carboplatin/cisplatin Q3w, for 4 cycles;JS004 200mg + JS001 240 mg + pemetrexed, maintained until disease progression
  Interventions: Biological: Recombinant humanized anti-BTLA monoclonal antibody (JS004) injection; Biological: Toripalimab; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin
- Cohort 4 (Experimental): NSCLC-squamous cell carcinoma first line;JS004 200mg + JS001 240 mg + paclitaxel + carboplatin Q3w, for 4 cycles; JS004 200mg + JS001 240 mg, maintained until disease progression
  Interventions: Biological: Recombinant humanized anti-BTLA monoclonal antibody (JS004) injection; Biological: Toripalimab; Drug: Carboplatin; Drug: Paclitaxel
- Cohort 5 (Experimental): SCLC first line;JS004 200mg + JS001 240 mg + etoposide + carboplatin/cisplatin Q3w, for 4 cycles; JS004 200mg + JS001 240 mg, maintained until disease progression
  Interventions: Biological: Recombinant humanized anti-BTLA monoclonal antibody (JS004) injection; Biological: Toripalimab; Drug: Cisplatin; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Biological: Recombinant humanized anti-BTLA monoclonal antibody (JS004) injection — 200mg via IV infusion once every 3 weeks;JS004 will be administered in combination with toripalimab until disease progression or intolerable toxicity or up to 2 years of treatment or other reasons specified in the protocol
Biological: Toripalimab — 240mg via IV infusion once every 3 weeks;JS004 will be administered in combination with toripalimab until disease progression or intolerable toxicity or up to 2 years of treatment or other reasons specified in the protocol
Drug: Docetaxel — 60 or 75mg/m2 via IV infusion on Day 1 of a 21-day cycle, which may be maintained until disease progression
  Arms: Cohort 2
Drug: Pemetrexed — 500mg/m2 via IV infusion on Day 1 of a 21-day cycle for 4 cycles; Subjects who have disease progression after 4 cycles may continue to receive maintenance treatment with pemetrexed
  Arms: Cohort 3
Drug: Cisplatin — 75mg/m2 via IV infusion on Day 1 of a 21-day cycle for 4 cycles
  Arms: Cohort 3; Cohort 5
Drug: Carboplatin — AUC 5 via IV infusion on Day 1 of a 21-day cycle for 4 cycles
  Arms: Cohort 3; Cohort 4; Cohort 5
Drug: Paclitaxel — 175mg/m2 via IV infusion on Day 1 of a 21-day cycle for 4 cycles
  Arms: Cohort 4
Drug: Etoposide — 100mg/m2 via IV infusion on Days 1, 2, and 3 of a 21-day cycle for 4 cycles
  Arms: Cohort 5

SUMMARY:
This is an open-label phase Ib/II clinical study to evaluate the safety, tolerability, pharmacokinetics and initial efficacy of JS004 injection combined with toripalimab and with or without standard chemotherapy in patients with advanced lung cancer

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible for the study if they meet all of the following criteria:

1. Sign the informed consent form voluntarily;
2. Males or females ≥18 years at the time of signing the informed consent;
3. Expected survival ≥3 months;
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 ;
5. Pathologically confirmed locally advanced, metastatic or recurrent non-small cell lung cancer (NSCLC), which is currently not suitable for local treatment such as radical surgery or radiotherapy; For subjects with non-squamous carcinoma, there is no EGFR sensitive mutation or ALK fusion; for subjects with squamous carcinoma, genetic testing is not mandatory
6. Pathologically confirmed extensive-stage small cell lung cancer (ES-SCLC, according to the Veterans Administration Lung Study Group (VALG) staging), previously received no systemic anti-tumor therapy for ES-SCLC (Cohort 5); Subjects with limited-stage SCLC who have previously received systemic anti-tumor therapy cannot be enrolled;
7. The subject has at least one measurable lesion as a target lesion (RECIST v1.1 criteria,);
8. The subject agrees to provide tumor tissue samples ;
9. The subject has good organ function as indicated by screening laboratory results:
10. Males of reproductive potential or females of childbearing potential must use effective contraceptive methods during the trial and continue for 6 months after the end of treatment;
11. The subject has good compliance and cooperates with the follow-up.

Exclusion Criteria:

Subjects who met any of the following criteria will be excluded from the study:

1. For the third line and second line populations with advanced lung squamous carcinoma (Cohorts 1 and 2), subjects who have received systemic anti-tumor therapy within 3 weeks before the first dose of study drug, including: chemotherapy, targeted therapy, anti-vascular drug therapy, biological therapy, immunotherapy, radiotherapy or other treatments with investigational products
2. Any adverse reactions caused by previous treatments have not recovered to CTCAE (Version 5.0) Grade 1 or below ;
3. Symptomatic metastases to central nervous system.;
4. Subjects with poorly controlled tumor-related pain who require analgesic treatment must receive the treatment at a stable dose before participating in the study;
5. Hydrothorax or ascites or pericardial effusion with clinical symptoms or unstable condition after symptomatic treatment;
6. Subjects previously discontinued treatment due to PD-1/PD-L1 inhibitor toxicity;
7. Known history of severe allergic reactions to JS004 or toripalimab and its components, scheduled chemotherapeutic drugs and their components;
8. Known active or suspected autoimmune diseases, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease;
9. History of interstitial lung disease or drug-induced interstitial lung disease or pulmonitis;
10. Received systemic corticosteroids (prednisone >10 mg/day or equivalent) or other immunosuppressive drugs within 14 days before the first study dose;
11. Subjects with a past history of immunodeficiency, including those with other acquired or congenital immunodeficiency diseases, or with a history of organ transplantation, or have received allogeneic hematopoietic stem cell transplantation or solid organ transplantation;
12. Had received live vaccines within 4 weeks before the first study dose;
13. Any major surgical procedure within 4 weeks before the first study dose. Planned major surgical procedure to be performed within 30 days after the first dose , or not fully recovered from the previous surgery;
14. Suffering from severe cardiovascular and cerebrovascular diseases;
15. Subjects with uncontrolled or serious underlying diseases, including but not limited to active infection requiring systemic antibiotic treatment;
16. Positive human immunodeficiency virus (HIV) antibody test, active hepatitis B or C;
17. Known active Pulmonary tuberculosis (TB)..
18. Any active malignancy other than the disease under study within the past 2 years, except for malignancies that can be expected to be cured after treatment;
19. Subjects who have a history of psychotropic drug abuse and are unable to withdraw or have mental disorder;
20. Pregnant or breastfeeding woman;
21. Other severe, acute or chronic medical or psychiatric disorders or laboratory abnormalities that, at the discretion of the investigator, may increase the risk associated with study participation or may interfere with the interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2025-10-23 (Actual); Study Completion 2025-10-23 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | 2 years
  Incidence of adverse events (AEs)
Incidence of SAEs | 2 years
  Incidence of serious adverse events (SAEs)
Incidence of irAEs | 2 years
  Incidence of immune-related adverse events (irAEs)
ORR | 2 years
  Efficacy endpoint: objective response rate (ORR) based on RECIST v1.1 criteria

SECONDARY OUTCOMES:
DOR | 2 years
  Efficacy endpoints: duration of response
DCR | 2 years
  Efficacy endpoints: disease control rate
time to response (TTR) | 2 years
  Efficacy endpoints: time to response
PFS | 2 years
  Efficacy endpoints: progression-free survival
OS | 2 years
  Efficacy endpoints: overall survival (OS)
1-year OS rate | 1 year
  Efficacy endpoints: 1-Year overall survival (OS) rate
Drug concentration in plasma | 2 years
  drug concentration at different time points after administration in an individual subject
incidence of ADA | 2 years
  incidence of anti-drug antibodies (ADA)
titer of ADA | 2 years
  titer of anti-drug antibodies (ADA)
incidence of Nab | 2 years
  incidence of neutralizing antibodies (Nab)
titer of Nab | 2 years
  titer of neutralizing antibodies (Nab)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No